CLINICAL TRIAL: NCT02220452
Title: The Effect of Intraoperative Music Listening on Sevoflurane Consumption and Recovery Parameters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Associate Professor in Anaesthesiology, Aretaieion University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Sofia-Music
Record Dates: First submitted 2014-08-17; First posted 2014-08-20 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Anesthesia; Stress; Music; Auditory Perception

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- music listening during anesthesia (Experimental): In patients allocated to the music listening group, audiotapes will be placed on patients' ears, playing soothing and relaxing music throughout anesthesia
  Interventions: Other: music listening during anesthesia
- absence of music listening during anesthesia (Active Comparator): In patients allocated to absence of music listening group, audiotapes will be placed on the patients' ears, without however playing any music
  Interventions: Other: absence of music listening during anesthesia

INTERVENTIONS:
Other: music listening during anesthesia — In patients allocated to the music listening group, audiotapes will be placed on patients' ears, playing soothing and relaxing music throughout anesthesia
  Arms: music listening during anesthesia
Other: absence of music listening during anesthesia — In patients allocated to absence of music listening group, audiotapes will be placed on the patients' ears, without however playing any music
  Arms: absence of music listening during anesthesia

SUMMARY:
* The perioperative period can be a significant source of psychological burden, anxiety and fear for patients
* Both pharmacological and non-pharmacological methods have been proposed in order to alleviate perioperative stress
* Music is one of the non-pharmacological methods which have been used in this context, with favorable effects both preoperatively and postoperatively
* The attenuation of perioperative stress through music listening is probably due to the activation of emotional and cognitive processes that evoke feeling of pleasure and can distract patients' attention from fear and unpleasant thoughts related to the surgical procedure
* Little information is available regarding the effect of intraoperative music listening on anesthetized, unconscious patients
* There is a notion that general anesthesia does not completely abolish auditory perception and that some processing of intraoperative events can occur in unconscious patients, even in the absence of postoperative recall
* The investigators hypothesis is that intraoperative music listening can decrease anesthetic requirements and reduce sevoflurane consumption in female patients subjected to abdominal hysterectomy for benign disease.

DETAILED DESCRIPTION:
* The perioperative period can be a significant source of psychological burden, anxiety and fear for patients
* Both pharmacological and non-pharmacological methods have been proposed in order to alleviate perioperative stress
* Music is one of the non-pharmacological methods which have been used in this context, with favorable effects both preoperatively and postoperatively
* Listening to music during the preoperative period has proved useful as an adjunct to premedication and can even be used instead of premedication. Additionally, listening to music postoperatively can also be useful, since it has been related to a more favorable recovery profile and possible attenuation of postoperative pain. In this context, music has also been used in Intensive Care Units, with measurable effects on anxiety scales and hemodynamic parameters. There are also studies investigating the use of music during operations under regional anesthesia, which have shown that music listening substantially decreases the need for anxiolytic administration throughout the operation
* The attenuation of perioperative stress through music listening is probably due to the activation of emotional and cognitive processes that evoke feelings of pleasure and can distract patients' attention from fear and unpleasant thoughts related to the surgical procedure
* Although the favorable effects of music listening during regional anesthesia for the attenuation of intraoperative stress in conscious patients are more or less expected and easily interpreted, less is known regarding the effect of intraoperative music listening on anesthetized, unconscious patients
* Generally, there is a notion that general anesthesia does not completely abolish auditory perception and that some processing of intraoperative events can occur in unconscious patients, even in the absence of postoperative recall
* The preservation of some form of auditory processing during general anesthesia is not necessarily undesirable and can be used to the patient's benefit, since it has been shown that subjecting patients to therapeutic suggestions during general anesthesia can improve recovery parameters or decrease hospital stay
* The investigators hypothesis is that intraoperative music listening can decrease anesthetic requirements. Therefore, the investigators will investigate sevoflurane consumption necessary to achieve a depth of anesthesia corresponding to bispectral index values of 45-55. Female patients subjected to abdominal hysterectomy for benign disease will be randomized to one of two groups: in the first group, audiotapes playing relaxing soothing orchestral music will be placed on the patients' ears after induction of general anesthesia while in the other group the same set of audiotapes will be used without however playing any music
* Sevoflurane consumption will be estimated by weighing the sevoflurane vaporizer in a high-precision scale before induction and after completion of the surgical procedure. Patients will also be queried regarding recall of any sounds or intraoperative events, dreaming while anesthetized and they will be asked to rate their satisfaction from anesthesia. Recovery parameters will also be investigated, such as postoperative nausea and vomiting and the intensity of postoperative pain. To ensure homogeneity, standardized analgesia will be administered in the two groups
* Since prolactin is related to the neuroendocrine response to stress, blood will also be sampled at predetermined timepoints during anesthesia, to detect potential differences between the two groups
* The clinical interest of this study lies in the fact that if a non-costly intervention such as music listening during anesthesia can lead to reduced requirements of anesthetic agents or to reduced need for postoperative analgesia, this theoretically can be translated to a reduction in anesthetic cost. In addition, improvement in recovery profile parameters could lead to a quicker discharge from the post-anesthesia care unit with reduction in turnaround times and overall time optimization.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, American Society of Anesthesiologists (ASA) distribution I-III, scheduled for elective hysterectomy for benign disease

Exclusion Criteria:

* hearing impairment
* psychiatric disease (depression, dementia)
* mental disability
* concurrent treatment with medication known to affect anesthetic requirement, such as benzodiazepines, anticonvulsants, opioids, psychotropic drugs or alcohol

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-08; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
sevoflurane consumption during general anesthesia | change of sevoflurane vaporizer weight from before induction to end of anesthesia, an average period of 2 hours
  the sevoflurane vaporizer will be weighed before anesthetic induction and at the end of anesthesia and consequently sevoflurane consumption during anesthesia will be determined

SECONDARY OUTCOMES:
recall of postoperative events | participants will be followed for the duration of stay in postanesthesia care unit, an average period of 1 hour
  a questionnaire will be used to assess the specific outcome measure
recall of postoperative sounds | participants will be followed for the duration of stay in postanesthesia care unit, an average period of 1 hour
  a questionnaire will be used to assess the specific outcome measure
occurence of postoperative nausea or vomiting | participants will be followed for the duration of stay in postanesthesia care unit, an average period of 1 hour
  a questionnaire will be used to assess the specific outcome measure
intensity of postoperative pain | participants will be followed for the duration of stay in postanesthesia care unit, an average period of 1 hour
  a verbal rating scale will be used to assess the specific outcome measure
satisfaction from anesthesia | participants will be followed for the duration of stay in postanesthesia care unit, an average period of 1 hour
  a verbal rating scale will be used to assess the specific outcome measure
measurement of prolactin levels | during the time that patients are anesthetized, an approximate period of 2 hours

OTHER OUTCOMES:
sleep diary | first postoperative night
  a questionnaire will be used to assess the specific outcome measure and participants will be queried in the first postoperative morning
sleep diary | second postoperative night
  a questionnaire will be used to assess the specific outcome measure and participants will be queried in the second postoperative morning

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, PhD, DEAA, Principal Investigator — Aretaieion University Hospital
Locations (1):
- Aretaieion University Hospital, Athens, Greece

REFERENCES:
- [Background] Bringman H, Giesecke K, Thorne A, Bringman S. Relaxing music as pre-medication before surgery: a randomised controlled trial. Acta Anaesthesiol Scand. 2009 Jul;53(6):759-64. doi: 10.1111/j.1399-6576.2009.01969.x. Epub 2009 Apr 14. PMID 19388893
- [Background] Wang SM, Kulkarni L, Dolev J, Kain ZN. Music and preoperative anxiety: a randomized, controlled study. Anesth Analg. 2002 Jun;94(6):1489-94, table of contents. doi: 10.1097/00000539-200206000-00021. PMID 12032013
- [Background] Ganidagli S, Cengiz M, Yanik M, Becerik C, Unal B. The effect of music on preoperative sedation and the bispectral index. Anesth Analg. 2005 Jul;101(1):103-6, table of contents. doi: 10.1213/01.ANE.0000150606.78987.3B. PMID 15976214
- [Background] Zhang XW, Fan Y, Manyande A, Tian YK, Yin P. Effects of music on target-controlled infusion of propofol requirements during combined spinal-epidural anaesthesia. Anaesthesia. 2005 Oct;60(10):990-4. doi: 10.1111/j.1365-2044.2005.04299.x. PMID 16179044
- [Background] Block RI, Ghoneim MM, Sum Ping ST, Ali MA. Human learning during general anaesthesia and surgery. Br J Anaesth. 1991 Feb;66(2):170-8. doi: 10.1093/bja/66.2.170. PMID 1817616
- [Background] Evans C, Richardson PH. Improved recovery and reduced postoperative stay after therapeutic suggestions during general anaesthesia. Lancet. 1988 Aug 27;2(8609):491-3. doi: 10.1016/s0140-6736(88)90131-6. PMID 2900410
- [Background] Lindh A, Carlstrom K, Eklund J, Wilking N. Serum steroids and prolactin during and after major surgical trauma. Acta Anaesthesiol Scand. 1992 Feb;36(2):119-24. doi: 10.1111/j.1399-6576.1992.tb03436.x. PMID 1532279